CLINICAL TRIAL: NCT04485832
Title: Telehealth Could Mitigate Disease Progression Compared to Standard of Care in COPD - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Frank Rassouli, PD Dr. med., Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BASEC Nr. 2015-00065
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Device: Telehealth care; Diagnostic Test: Weekly CAT measurement
- Control (Active Comparator)
  Interventions: Diagnostic Test: Weekly CAT measurement

INTERVENTIONS:
Device: Telehealth care — Patients in the intervention group daily answer 6 questions, which are focused on the recognition of AECOPD, using the electronic healthcare platform Evita by Swisscom, which has been and continuously is developed by the study team and Swisscom. The study team daily analyses all patients online and reacts according to a pre-specified action plan.
  Arms: Intervention
Diagnostic Test: Weekly CAT measurement

SUMMARY:
The objective of this randomised controlled trial is to test, whether telehealthcare can improve HRQOL and reduce emergency admissions and hospitalisations due to AECOPD. Different outcome parameters as described in the endpoints section will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD B-D and age ≥ 40 years

Exclusion Criteria:

* Inability to provide informed consent or to follow trial procedures

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change of COPD assessment test (CAT) at 6 months (slope of the linear regression trend) | 1 year after inclusion

IPD SHARING:
Plan to Share IPD: No